CLINICAL TRIAL: NCT04181060
Title: Randomized Phase III Study of Combination Osimertinib (AZD9291) and Bevacizumab Versus Osimertinib (AZD9291) Alone as First-Line Treatment for Patients With Metastatic EGFR-Mutant Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Osimertinib With or Without Bevacizumab as Initial Treatment for Patients With EGFR-Mutant Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-07941; NCI-2019-07941 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA5182 (Other: ECOG-ACRIN Cancer Research Group); EA5182 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2019-11-27; First posted 2019-11-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lung Non-Squamous Non-Small Cell Carcinoma; Metastatic Lung Non-Squamous Non-Small Cell Carcinoma; Recurrent Lung Non-Squamous Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Magnetic Resonance Spectroscopy; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (osimertinib) (Active Comparator): Patients receive osimertinib PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO, MUGA, CT and may undergo MRI and blood and urine sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Osimertinib
- Arm B (osimertinib, bevacizumab) (Experimental): Patients receive osimertinib PO QD on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO, MUGA, CT and may undergo MRI and blood and urine sample collection on study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Osimertinib

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm B (osimertinib, bevacizumab)
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib

SUMMARY:
This phase III trial compares the effect of bevacizumab and osimertinib combination vs. osimertinib alone for the treatment of non-small cell lung cancer that has spread outside of the lungs (stage IIIB-IV) and has a change (mutation) in a gene called EGFR. The EGFR protein is involved in cell signaling pathways that control cell division and survival. Sometimes, mutations in the EGFR gene cause EGFR proteins to be made in higher than normal amounts on some types of cancer cells. This causes cancer cells to divide more rapidly. Osimertinib may stop the growth of tumor cells by blocking EGFR that is needed for cell growth in this type of cancer. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Giving osimertinib with bevacizumab may control cancer for longer and help patients live longer as compared to osimertinib alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate progression-free survival (PFS) of osimertinib (AZD9291) and bevacizumab versus osimertinib (AZD9291) alone as first-line treatment for patients with metastatic EGFR-mutant lung cancers.

SECONDARY OBJECTIVES:

I. To evaluate overall survival (OS). II. To evaluate best objective response rate and duration of objective response.

III. To evaluate time to central nervous system (CNS) progression and CNS PFS. IV. To evaluate toxicity of the combination regimen.

CORRELATIVE OBJECTIVES:

I. To characterize mechanisms of resistance to osimertinib (AZD9291) and osimertinib (AZD9291) with bevacizumab first-line therapy through post-progression circulating tumor-derived deoxyribonucleic acid (ctDNA).

II. To assess for ctDNA clearance on study treatment and associate ctDNA clearance with clinical outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive osimertinib orally (PO) once daily (QD) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive osimertinib PO QD on days 1-21 and bevacizumab intravenously (IV) over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo echocardiography (ECHO), multigated acquisition scan (MUGA), computed tomography (CT) and may undergo magnetic resonance imaging (MRI) and blood and urine sample collection on study.

After completion of study treatment, patients are followed up every 3 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a pathologically-confirmed diagnosis of non-squamous, non-small cell lung cancer (NSCLC)
* Patient must have advanced disease, defined as - either stage IV disease, stage IIIB disease not amenable to definitive multi-modality therapy, or recurrent disease after a prior diagnosis of stage I-III disease. All staging is via the American Joint Committee on Cancer (AJCC)/International Association for the Study of Lung Cancer (IASLC) 8th edition staging criteria
* Patient must have somatic activating sensitizing mutation in EGFR (e.g. but not limited to Exon 19 deletion, L858R, E709X, G719X, exon 19 insertions, L861Q, S768I). Patients with non-sensitizing mutations in EGFR (EGFR exon 20 insertions) are not eligible. Test results originating from a Clinical Laboratory Improvement Act (CLIA)-certified or similarly accredited laboratory are acceptable; no specific assay is mandated. Plasma, cytology, or tumor tissue can be utilized for mutation testing
* Patient must not have received any prior treatment with an anti-VEGF agent

  * NOTE: Prior treatment with an EGFR TKI is not allowed, however if a candidate for this study has already started osimertinib within 21 days prior to randomization, the exact osimertinib start date is known, and the patient had the required study baseline imaging completed prior to the osimertinib start date, the patient will be eligible
* Patients that have received prior radiation therapy are eligible. Radiation (limited field stereotactic radiation or conventional radiation) must have been completed at least one week prior to study drug initiation and more extensive field radiation (i.e., whole-brain radiotherapy [WBRT]) must have been completed at least two weeks prior to drug initiation
* Patient must not have any risk factors for anti-VEGF administration, specifically, hemoptysis, active cardiovascular disease, uncontrolled hypertension, significant proteinuria (screening urinalysis > 300 mg/dl) and tumor invading major blood vessels
* Patient must have measurable disease. Baseline measurements of sites of disease must be obtained within 4 weeks prior to study randomization. If a potential target lesion is previously irradiated without subsequent growth and/or is radiated after the imaging from which baseline measurements are obtained, they cannot be included as target lesions, and additional target lesions are required to meet criteria for measurable disease
* Patient must not have had any prior systemic treatment for metastatic disease
* Patient must be ≥ 18 years of age
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used
* All females of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy
* A female of childbearing potential is defined as any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient of childbearing potential and sexually active males must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for 2 weeks prior to the start of treatment, while on study treatment, and for

  * 6 weeks after the last dose of protocol treatment for female patients on the osimertinib (AZD9291) alone arm
  * 4 months after the last dose of protocol treatment for male patients on osimertinib (AZD9291) alone arm
  * 6 months after the last dose of protocol treatment for all patients on osimertinib (AZD9291) plus bevacizumab combination arm
  * NOTE: Female patients should also not breastfeed while on treatment and for 6 months after the last dose bevacizumab
* Leukocytes >= 3,000/mcL (obtained =< 14 days prior to randomization)
* Absolute neutrophil count >= 1,500/mcL (obtained =< 14 days prior to randomization)
* Platelets >= 100,000/mcL (obtained =< 14 days prior to randomization)
* Hemoglobin >= 9 g/dL (obtained =< 14 days prior to randomization)
* Total bilirubin and creatinine =< 1.5 x institutional upper limit of normal (ULN) (obtained =< 14 days prior to randomization)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (obtained =< 14 days prior to randomization)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if neurologically stable without glucocorticoid therapy after the stated washout period from radiation therapy (RT) or surgery provided the metastatic lesions are non-hemorrhagic
* Patients with untreated brain metastases or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required provided the metastatic lesions are non-hemorrhagic and are neurologically stable without glucocorticoid therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patient must have the ability to understand and the willingness to sign a written informed consent document and comply with study requirements
* Patient must not have had treatment with any investigational drug within five half-lives or 3 months (whichever is greater), prior to study initiation
* Patient must not be currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4. For any patient currently receiving such inducers of CYP3A4, they must discontinue use prior to first dose of study treatment. All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4
* Patient must not have any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of randomization, with the exception of alopecia and grade 2 prior platinum-therapy-related neuropathy
* Patient must not have any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it challenging for the patient to participate in the study. Screening for chronic conditions is not required
* Patient must not have refractory nausea and vomiting, chronic gastrointestinal diseases, the inability to swallow the osimertinib tablets or previous significant bowel resection that would preclude adequate absorption of osimertinib
* Patient must not have a medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* Patient must not have a history of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib
* Patient must not have mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value (using Bazett's correction)
* Patient must not have any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second-degree heart block
* Patient must not have any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: potassium < lower limit of normal [LLN]; magnesium < LLN; calcium < LLN), congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause torsades de pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to documented disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or death from any cause, whichever occurs first, assessed up to 10 years
  Will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate the treatment hazard ratios. PFS will use a logrank test stratified on the randomization stratification factors with a one-sided type I error rate of 2.5%.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, assessed up to 10 years
  Will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate the treatment hazard ratios. OS will be tested at the one-sided 10% level.
Best objective response rate | Up to 10 years
  Best objective response will be evaluated via RECIST 1.1 criteria. Will be compared using Fisher's exact tests with a one-sided type I error rate of 2.5%; multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes.
Time to central nervous system progression | From study randomization to evidence of central nervous system progressive disease, with death and progression as competing events, assessed up to 10 years
  Will be estimated using competing risks methodology, adjusting for death and progression as competing events. Regular central nervous system imaging will occur when patients are on treatment. After they discontinue study treatment, central nervous system imaging will be symptom-prompted during follow up.
Central nervous system progression-free survival | From study randomization to evidence of central nervous system progressive disease or death from any cause, whichever occurs first, assessed up to 10 years
  Will be estimated using the Kaplan-Meier method.
Incidence of adverse events | Up to 30 days after the last administration of investigational agent
  Toxicity will be determined using the Common Terminology Criteria for Adverse Events (CTCAE). Will be compared using Fisher's exact tests with a one-sided type I error rate of 2.5%; multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes.

OTHER OUTCOMES:
Mechanisms of resistance to AZD9291 (osimertinib) and AZD9291 (osimertinib) with bevacizumab first-line therapy through post-progression circulating tumor-derived deoxyribonucleic acid (ctDNA) | Up to 10 years
  Preliminary analyses of these data will utilize tests for association comparing the frequency of a particular genomic aberration at baseline and at progression (for example, using McNemar's test) and association between alterations and baseline characteristics (for example, using Fisher's exact test). More sophisticated analyses may include multivariable logistic regression modeling and/or competing risks analysis.
Circulating tumor deoxyribonucleic acid (ctDNA) clearance on study treatment | Up to 10 years
  Will assess ctDNA clearance on study treatment and associate ctDNA clearance with clinical outcomes. Cox regression analysis will be used to assess whether EGFR ctDNA clearance is an independent predictor for PFS (and OS), adjusted by treatment effect, the presence of brain metastasis (yes versus [vs.] no), EGFR exon 19 deletion/L858R vs other, Eastern Cooperative Oncology Group (ECOG) performance status (0-1 vs 2) and other possible clinical and biological risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Helena A Yu, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (603):
- United States (603):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Houston Methodist Cypress Hospital, Cypress, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm